CLINICAL TRIAL: NCT04439916
Title: Breakthrough CMV DNAemia in CMV Seronegative Recipients of CMV Seropositive Lung Transplantation During Antiviral Prophylaxis With Valganciclovir. A Pilot Study.
Brief Title: Breakthrough CMV Lung Transplant -Multicentre
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00093295
Record Dates: First submitted 2020-06-08; First posted 2020-06-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cytomegalovirus Infections
Keywords: CMV; Lung transplant; Valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cytomegalovirus (CMV) infection is the most common opportunistic infection in lung transplantation leading to direct and indirect effects that can result in life threatening complications. The risk of CMV infection is highest when the recipient of the transplant has never been in contact with CMV (negative immunity) and the donor had previous contact with CMV (positive immunity). This is called CMV mismatch. For these lung transplant patients 6 to 12 months of prophylaxis with an antiviral called Valganciclovir is recommended. This antiviral can cause side effects like bone marrow toxicity and decrease in immune cells which can result in temporarily having to stop the treatment. Starting and stopping the prophylaxis may result in the CMV becoming resistant to the medication. While taking the prophylaxis it is possible to have a breakthrough of the CMV, this is often due to the development of resistance to the antiviral. The purpose of this study is to learn more about the rate of CMV breakthrough while on prophylaxis after lung transplantation in patients who are CMV mismatch. The investigators will also look at the rates of negative side effects caused by antiviral prophylaxis in this population.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to learn more about the rate of CMV breakthrough in lung transplant patients who are CMV mismatched and receiving prophylaxis. The rates of negative side effects caused by the antiviral prophylaxis will also be monitored. For patients who do have a breakthrough of CMV viremia while on study the investigator will also evaluate the rate of resistance mutations.

Hypothesis:

The investigator wants to demonstrate that breakthrough CMV DNAemia is common in CMV mismatch lung transplant recipients on ganciclovir/valganciclovir prophylaxis. In addition, the investigator will show that leukopenia and neutropenia related to prolonged prophylaxis is very common and discontinuation of ganciclovir/valganciclovir prophylaxis because of side effects explains most cases of breakthrough CMV DNAemia. The investigators findings will be relevant because they will answer the following questions:

1. Prophylaxis with ganciclovir/valganciclovir in mismatch lung transplant patients should include intensive CMV DNA monitoring.
2. Side effects related to the use of ganciclovir/valganciclovir can result in potential life-threatening infections due to the development of neutropenia and increased cost due to the use of granulocyte-colony stimulating factor.
3. Alternative prophylaxis with new antivirals with safer profile of side effects would result in a safer profile of adverse events. As resistance to ganciclovir may lead to death, the development of CMV infection in patients receiving antivirals targeting different enzymes than those targeted by ganciclovir/valganciclovir will not prevent future use of ganciclovir/valganciclovir to treat CMV infection or disease.

Justification:

Cytomegalovirus (CMV) infection is the most common opportunistic infection in lung transplantation leading to direct and indirect effects that can result in life threatening complications. The risk of CMV infection is highest in CMV seronegative lung recipients from CMV seropositive donor (CMV mismatch). Antiviral prophylaxis for 6 to12 months with valganciclovir is indicated in CMV mismatch lung transplant recipients according to International Guidelines. Despite prolonged antiviral prophylaxis, the risk of CMV infection post-prophylaxis is high in this group of patients. Valganciclovir was approved for antiviral prophylaxis in organ transplant patients in 2004. Rates of breakthrough CMV infection may be higher after 6 months of prophylaxis due to an increased risk of bone marrow toxicity and neutropenia from Valganciclovir that may lead to temporary prophylaxis discontinuation.

Resistance to ganciclovir is a major complication in all solid organ transplant patients, but lung transplant recipients are the subgroup of patients at highest risk. The rate of ganciclovir-resistant CMV infection in CMV mismatch lung transplant recipients is the highest among all organ transplants and its occurrence is associated with increased risk of death. Although CMV mismatch lung transplantation has been found to be a risk factor for ganciclovir-resistant CMV infection in most of the studies, the underlying pathophysiological mechanisms are not fully understood. Discontinuation of valganciclovir can lead to CMV replication with exposure to sub-therapeutic levels of ganciclovir in blood, and this may lead to the development of antiviral resistance.

Objectives:

1. To evaluate the incidence of breakthrough CMV infection in CMV mismatch lung transplant patients receiving 6-12 months antiviral prophylaxis with ganciclovir/valganciclovir.
2. To evaluate the rates of leukopenia, neutropenia and antiviral prophylaxis discontinuation due to side effects of antiviral prophylaxis with ganciclovir/valganciclovir in CMV mismatch lung transplant patients.
3. To evaluate the rates of ganciclovir/valganciclovir resistance mutations in CMV DNA from mismatch lung transplant patients with breakthrough CMV viremia.

Research Method/Procedures:

This will be a prospective, multicenter, non-randomized, non-interventional study in 40 CMV mismatch lung transplant patients receiving standard of care prophylaxis according to each center. At baseline the patients medical history will be reviewed with them. Post transplant weeks 1 to 24 or 52 a CMV Polymerase chain reaction (PCR) will be done every two weeks. Standard of care blood work and the patients chart will be monitored to look for any relevant side effects or changes in medication. In case CMV viremia is detected during prophylaxis, the local PI can decide either to treat the CMV infection with therapeutic dose of antivirals (ganciclovir, valganciclovir or Foscarnet) or to maintain prophylaxis and CMV PCR monitoring. In all cases of CMV breakthrough viremia, a whole blood or plasma sample will be sent to Provincial Microbiology Lab in Edmonton to perform antiviral resistance by next-generation sequencing. From post transplant weeks 24 to 36 or 52 to 64 weekly CMV PCR will be done as per standard of care, all other standard of care blood work will also be monitored. Chart reviews will be completed to look for any relevant side effects.

Plan for Data Analysis:

For the analysis of data the investigator will have the support of the Northern Alberta Clinical Trials and Research Centre (NACTRC). Incidence rate of breakthrough CMV viremia, leukopenia, neutropenia and severe neutropenia will be calculated as number of case per 1,000 patients/week. The percentage of CMV infection post-prophylaxis in patients with and without breakthrough CMV infection will be compared by Fisher's exact test. Cox-regression analysis will be performed to identify independent variables associated with CMV breakthrough viremia.

ELIGIBILITY:
Inclusion Criteria:

* CMV seronegative recipients of CMV seropositive donor lung transplantation.
* Age 18 years or older.
* Receipt of antiviral prophylaxis with valganciclovir as per local protocol with a duration of 6 or 12 months after transplantation.
* Monitoring of CMV DNAemia post-prophylaxis for at least 12 weeks as per local protocol.
* Signed informed consent.

Exclusion Criteria:

* Known allergy to ganciclovir or valganciclovir.
* Neutropenia (< 1.0) pre-transplantation.
* Living-donor lung transplantation.
* Lung re-transplantation.
* Pre-transplant immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients, 18 years or older, who will receive either 6 or 12 months of prophylaxis, are CMV seronegative and received a CMV seropositive transplant.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CMV Breakthrough | Up to 52 weeks
  Incidence of CMV infection (defined as any quantifiable CMV viral load in plasma or blood) during prophylaxis. Will be categorized as CMV asymptomatic infection or CMV disease.

SECONDARY OUTCOMES:
CMV infection | 12 weeks
  Incidence of CMV infection post-prophylaxis (categorized as CMV infection or disease).
Neutropenia | through study completion, up to 64 weeks
  Absolute neutrophil count < 1,000 cells/mL
Severe neutropenia | through study completion, up to 64 weeks
  Absolute neutrophil count < 500 cells/mL
Leukopenia | through study completion, up to 64 weeks
  White cell count < 2,000 cells/mL
Use of Granulocyte - colony stimulating factor (G-CSF) | through study completion up, to 64 weeks
  Whether a patient requires G-CSF
CMV resistant infection | through study completion, up to 64 weeks
  Mutation in UL97, UL54 or both.
Opportunistic and non-opportunistic infections | through study completion, up to 64 weeks
  All incidence of other infections
Chronic lung allograft dysfunction | through study completion, up to 64 weeks
  All incidence of chronic lung allograft dysfunction will be captured.
Retransplantation | through study completion, up to 64 weeks
  Any incidence where retransplantation is required
Death | through study completion, up to 64 weeks
  Whether a patient dies during study

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Carlos Cervera, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada